CLINICAL TRIAL: NCT02806245
Title: Biventricular Pacing in Children After Surgery for Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Friedberg, Associate Scientist, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000010911
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Congenital Heart Disease (CHD); Cardiopulmonary Bypass (CPB); Cardiac Index; Hemodynamics; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biventricular pacing (Experimental): Patients will be randomized pre-operatively to either the pacing group or to the control group. Patients randomized to receive pacing will 1st undergo an acute pacing phase where the order of the pacing mode will be randomized and then will continue to an extended pacing phase of biventricular pacing.
  Interventions: Other: Biventricular pacing
- Control (No Intervention): Controls will receive standard of care treatment consisting of placement of 2 pacing leads (right atrial and right ventricular), monitoring of the study outcomes, monitoring of oxygen consumption and echocardiography, but no pacing.

INTERVENTIONS:
Other: Biventricular pacing — Randomization into one of 3 study arms for acute phase and for extended phase.
  Measurement of baseline variables on arrival to CCU. Acute pacing protocol (order of pacing randomized):
  1. Atrial sensing- right ventricular pacing 10 min.
  2. 5 min no pacing (washout).
  3. Atrial sensing - biventricular pacing 10 min.
  4. 5 min no pacing (washout).
  5. Intrinsic rhythm
  6. 5 min no pacing (washout). Start extended phase pacing according to randomization. Measure hemodynamic variables 10 min after start of pacing.
  Measure hemodynamic variables 30 min after start of pacing. Pacing hiatus for 60 minutes at 24 hours with measurement of hemodynamics without pacing and after reinitiating pacing.
  Stop pacing at 72 hours or after extubation, whichever comes first. For those patients who are extubated before 72 hours: measurements will be taken before extubation and one hour after extubation. Pacing will then be stopped.
  Arms: Biventricular pacing

SUMMARY:
Surgery with cardiopulmonary bypass (CPB) for congenital heart disease (CHD) causes low cardiac index (CI). With the increasing success of surgery for CHD, mortality has decreased and emphasis has shifted to post-operative morbidity and recovery. Children with CHD undergoing surgery with CPB can experience well-characterized post-operative cardiac dysfunction. When severe, patients can develop clinically important low cardiac output syndrome (LCOS) and hemodynamic instability. Management of LCOS and hemodynamic compromise is primarily accomplished via intravenous durgs like milrinone, dopamine or dobutamine, which affect the strength of the heart's muscular contractions. These are used to maintain adequate blood pressure (BP) and CI. However, inotropic agents are potentially detrimental to myocardial function and may increase risk for post-operative arrhythmia and impair post-operative recovery by increasing oxygen demand and myocardial oxygen consumption (VO2). In combination with the increased VO2 associated with CPB-induced systemic inflammatory response patients can develop a critical mismatch between oxygen supply and demand, essentially the definition of LCOS. Therefore, therapies that improve CI and hemodynamic stability without increased VO2 are beneficial. This study will test whether BiVp, a specialized yet simple pacing technique, can improve post-operative CI and recovery in infants with electro-mechanical dyssynchrony (EMD) after CHD surgery. This study hypothesizes that Continuous BiVp increases the mean change in CI from baseline to 72 hours in infants with EMD following CHD surgery compared to standard care alone.

DETAILED DESCRIPTION:
In adults with heart failure with intrinsic or iatrogenic left bundle branch block (eg, RV pacing), and more recently in those with narrow QRS complex, pacing the heart with advanced pacing techniques from both the left and right ventricle (LV, RV) termed cardiac resynchronization therapy (CRT) improves resting systolic heart function and mechanoenergetics.1 In these patients, CRT has been shown to increase LV stroke volume, ejection fraction, and stroke work, resulting in an enhancement of LV myocardial efficiency, without an increase in oxidative metabolism and even a decrease in energy utilization.2-4 Furthermore, oxygen consumption seems to be distributed more homogeneously during CRT.2 Beyond increasing resting myocardial efficiency, CRT may increase metabolic reserve as judged by the increase in cardiac work in response to dobutamine.5 CRT has also been shown to restore homogeneous myocardial glucose metabolism, without a decrease in myocardial perfusion.6 These findings were mirrored by similar findings regarding the effects of CRT on myocardial perfusion. Resting myocardial blood perfusion was unaltered by CRT despite an increase in left ventricular function. However, the distribution pattern of resting myocardial blood perfusion became more homogeneous, while hyperemic myocardial blood perfusion and myocardial blood perfusion reserve were enhanced by CRT.7 In the long-term, CRT improves morbidity and mortality in adults with heart failure.8, 9

Children have myocardial dysfunction and possibly mechanical dyssynchrony following cardiopulmonary bypass and cardiac surgery. A significant number of children with congenital heart disease have either interventricular conduction delay or right bundle branch block (RBBB). For example, RBBB may occur in patients after ventricular septal defect repair. Others children may develop iatrogenic bundle branch block while requiring ventricular pacing for rate control, hemodynamic improvement or atrioventricular block. When postoperative pacing is indicated, the current method used is to sense or pace the right atrium, depending on the indication, and to pace the right ventricle (univentricular pacing). However, conventional RV univentricular pacing may increase myocardial stress and oxygen utilization through inhomogeneous contraction,10 while long-term right ventricular (univentricular) pacing has been shown in some patients to have detrimental effects on left ventricular remodeling, left ventricular function and clinical outcomes.11-13 Beyond the potential for pacing related myocardial stress and oxygen consumption, the post-operative care of children with congenital heart disease necessitates the use of potent inotropic agents at the expense of increased myocardial oxygen consumption, unwanted effects in the vulnerable post-bypass myocardium.14-16 Preliminary data in children with congenital heart disease undergoing surgical repair have shown acute benefits of CRT as manifested by increased systolic blood pressure and improved cardiac output associated with a reduced QRS duration. These beneficial effects were obtained in children with both single and dual ventricular physiology.17-20 Pham et al showed improvement in cardiac index with biventricular pacing in children after heart surgery, but not with conventional atrioventricular pacing, suggesting that in patients needing pacing in the postoperative period, biventricular pacing is better than conventional pacing, a conclusion previously reached in adults in the setting of cardiomyopathy.21-23 Despite these beneficial immediate hemodynamic effects, and despite preliminary data on the beneficial effects of CRT in children with congenital heart disease,24-26 it is not known whether a longer period of biventricular pacing in the post-operative period following surgery for congenital heart disease is beneficial and whether this intervention can lead to improved clinical outcomes such as reduction of the use of inotropes, time to extubation and length of admission to the critical care unit. To answer these questions, a prospective, randomized trial is needed. The current study would serve as a pilot study for a larger trial in the event of encouraging results.

Hypothesis

Biventricular pacing improves recovery after cardiac surgery with cardiopulmonary bypass in children with congenital heart disease.

Objectives

Study the effects of biventricular pacing on post-operative hemodynamics and clinical outcomes in children after surgery for congenital heart disease.

Design

Randomized, non-blinded, clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* < 4 months of age at time of surgery
* Surgery for congenital heart disease requiring cardiopulmonary bypass
* Reparative surgery to achieve biventricular cardiac physiology.
* Sinus rhythm.

Exclusion Criteria:

* Isolated atrial septal defect repair.
* Surgery without cardiopulmonary bypass.
* Palliative surgery.
* Single ventricle physiology.
* Age > 4 months at time of surgery
* Clinical indication for pacing (e.g. iatrogenic heart block)
* Arrhythmia
* Second or third degree heart block.
* Patient with known bleeding disorder
* Patient requires ECMO in operating room (eg. unable to wean from cardio-pulmonary bypass or hemodynamic/ respiratory instability that requires ECMO in OR). These patients return from the OR to the ICU on ECMO.

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in mean cardiac index | Baseline to 72 hours
  1. Change in mean cardiac index (as measured by the Fick method with respiratory mass spectroscopy for VO2) from baseline to 48 postoperative hours after arrival in the CCCU, recorded every 6 hours up to 72 hours and at each time blood gases sampled.

SECONDARY OUTCOMES:
Composite clinical score | Baseline to 72 hours
  a.Time until first negative fluid balance b.Time until sternal closure c.Time until first planned extubation d.In-hospital death e.Extracorporeal membrane oxygenation
Oxygen consumption | Every hour for 1st 24 hrs and then every 6hours
  2. Oxygen consumption (respiratory mass spectroscopy), measured continuously, recorded every hour for the 1st 24 hours, then every 6 hours and at each blood gas sampling.
Intracardiac pressures (RA, LA, CVP, PA) | Every hour for the 1st 24 hours, then every 6 hours until lines removed
  Intracardiac pressures (RA, LA, CVP, PA) measured continuously, recorded every hour for the 1st 24 hours, then every 6 hours until lines removed.
Mean inotrope score | every hour for the 1st 24 hours, then every 6 hours
  Mean inotrope score recorded every hour for the 1st 24 hours, then every 6 hours.
Mean airway pressure | every hour for the 1st 24 hours, then every 6 hours
  Mean airway pressure recorded every hour for the 1st 24 hours, then every 6 hours (simultaneously with inotrope score)
Serum Lactate | Over 72 hours recorded every 6 hours
  Serum lactate over 72 hours, recorded every 6 hours.
Blood pressure | over 72 hours, recorded every hour for the 1st 24 hours and then every 6hours
  Blood pressure over 72 hours, recorded every hour for the 1st 24 hours and then every 6 hours
Length of stay in CCCU | Over 72 hours
  Length of stay in CCCU (recorded in hours).
Electrical dyssynchrony | Baseline and 48 hours
  Electrical dyssynchrony at 48 hours (QRS duration in msec from 6-lead limb ECG).
Echocardiograms | Baseline and 48 hours
  Echocardiograms will be done at baseline (after arrival in CCCU, before pacing) and at 48 hours after arrival to the CCCU to assess mechanical dyssynchrony.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Friedberg, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Friedberg MK, Schwartz SM, Zhang H, Chiu-Man C, Manlhiot C, Ilina MV, Arsdell GV, Kirsh JA, McCrindle BW, Stephenson EA. Hemodynamic effects of sustained postoperative cardiac resynchronization therapy in infants after repair of congenital heart disease: Results of a randomized clinical trial. Heart Rhythm. 2017 Feb;14(2):240-247. doi: 10.1016/j.hrthm.2016.09.025. Epub 2016 Sep 26. PMID 27687644